CLINICAL TRIAL: NCT05663593
Title: A Randomised, Double-blind, Placebo-controlled, 2-part Study to Assess the Safety, Tolerability, Pharmacokinetics, Pharmacodynamics and Food Effect of Single and Multiple Oral Doses of HSK31858 in Healthy Volunteers
Brief Title: Safety, Tolerability,PK/PD, Food Effect of Single and Multiple Ascending Doses of HSK31858 in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Haisco Pharmaceutical Group Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: HSK31858-102
Record Dates: First submitted 2022-12-06; First posted 2022-12-23 (Actual); Last update posted 2022-12-23 (Actual); Status verified 2022-09

CONDITIONS: Healthy Volunteers
Keywords: HSK31858; NCFBE; phase I
MeSH Terms: interventions — Tablets

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- HSK31858 (Experimental): Single or multiple oral doses of HSK31858 Tablet, orally once daily
  Interventions: Drug: HSK31858, tablet
- Placebo (Placebo Comparator): Matching placebo Tablet, orally once daily
  Interventions: Drug: Placebo, tablet

INTERVENTIONS:
Drug: HSK31858, tablet — Starting dose in single ascending dose: 5 mg
  Arms: HSK31858
Drug: Placebo, tablet — Matching placebo
  Arms: Placebo

SUMMARY:
This is a phase I, randomised, double-blind placebo-controlled, 2-part study to assess the safety, tolerability, pharmacokinetics, pharmacodynamics and food effect of single and multiple oral doses of HSK31858 in healthy volunteers

ELIGIBILITY:
Inclusion Criteria:

1. Must have given written informed consent before any study-related activities are carried out and must be able to understand the full nature and purpose of the trial, including possible risks and adverse effects.
2. Adult males and females, 18 to 45 years of age (inclusive) at Screening.
3. Body mass index ≥ 18.0 and ≤ 28.0 kg/m2, with a body weight ≥ 45 kg at Screening.
4. Be nonsmokers (including tobacco, e-cigarettes, and marijuana) for at least 1 month prior to first study drug administration.
5. Medically healthy without clinically significant abnormalities at Screening and predose on Day 1.
6. Conventional 12-lead ECG recording in triplicate (the mean of triplicate measurements will be used to determine eligibility at Screening and predose on Day 1) consistent with normal cardiac conduction and function.

Exclusion Criteria:

1. History or presence of significant cardiovascular, pulmonary, hepatic, renal, hematological, gastrointestinal, endocrine, immunologic, dermatologic or neurological disease, including any acute illness or surgery within the past 3 months determined by the PI to be clinically relevant.
2. Subjects has increased risk of infection:

   1. History and/or presence of tuberculosis (TB).
   2. Body temperature of > 37.7℃.
   3. Blood neutrophil count <1.5 × 109/L, or white blood cell count <3.5×109/L (Screening and Day -1).
   4. Is in high risk-group (i.e., men who have had unprotected sex with men, women who have had sex without a condom with men who have sex with men, people who have had sex without a condom with a person who has lived or travelled in Africa, people who inject drugs, people who have had sex without a condom with somebody who has injected drugs, people who have caught another sexually transmitted infection, people who have received a blood transfusion while in Africa, eastern Europe, the countries of the former Soviet Union, Asia or central and southern America) for human immunodeficiency virus (HIV) infection within the last 6 months.
   5. Other latent or chronic infections (e.g., recurrent sinusitis, genital or ocular herpes, urinary tract infection) or at risk of infection (surgery, trauma, or significant infection) within 3 months of Screening, or history of skin abscesses within 3 months of Screening.
   6. Clinically significant lower respiratory tract infection not resolved within 4weeks prior to Screening, as determined by the PI.
   7. Volunteers with active malignancy or neoplastic disease in the previous 5 years other than superficial basal cell carcinoma.
   8. Disease history suggesting abnormal immune function or use of or plans to use systemic immunosuppressive (e.g., corticosteroids, methotrexate, azathioprine, cyclosporine) or immunomodulating medications (e.g., interferon) during the study or within 4 months prior to the first study drug administration.
3. Some subjects lacking functional Dipeptidyl peptidase 1 (DPP1) enzyme have been described to have periodontitis and palmoplantar hyperkeratosis:

   1. Subjects with signs of current gingivitis/periodontitis. Gingival evaluation (by inspection) will be performed by a dental hygienist or trained study physician.
   2. Subjects with a history of hyperkeratosis or erythema in palms or soles.
4. Liver function test results (i.e., aspartate aminotransferase [AST], alanine aminotransferase [ALT], and gamma glutamyl transferase [GGT]) and total bilirubin elevated more than 1.5 fold above the ULN.
5. Hepatitis B surface antigen (HBsAg), hepatitis C antibody (HCVAb), syphilis antibody and human immunodeficiency virus (HIV) antibody test are positive at screening.
6. Presence or having sequelae of gastrointestinal, liver, kidney, or other conditions known to interfere with the absorption, distribution, metabolism, or excretion of drugs.
7. History of alcohol abuse within 12 months prior to first study drug administration or positive alcohol breath test. Regular alcohol consumption defined as > 21 alcohol units per week (where 1 unit = 284 mL of beer, 25 mL of 40% spirit or a 125 mL glass of wine).
8. Use of any prescription or over-the-counter medication (including herbal products, diet aids, and hormone supplements) within 14 days or 5 half-lives of the medication (whichever is longer) prior to the first study drug administration, except occasional use of paracetamol. Use of any IP or investigational medical device within 30 days prior to Screening, or 5 half-lives of the product (whichever is the longest).
9. Donation of blood or plasma within 30 days prior to first study drug administration, or loss of whole blood of more than 500 mL within 30 days prior to randomization, or receipt of a blood transfusion within 1 year of first study drug administration.
10. Participation in another investigational clinical trial within 60 days prior to the first study drug administration.

19. Pregnant or lactating at Screening or planning to become pregnant (self or partner) at any time during the study, including the Follow-up period.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 74 (Actual)
Dates: Start 2022-02-23 (Actual); Primary Completion 2022-08-15 (Actual); Study Completion 2022-11-30 (Actual)

PRIMARY OUTCOMES:
The number and severity of treatment emergent adverse events (TEAEs) | 7 days after single dose
  To assess the safety and tolerability of single oral dose of HSK31858 in healthy volunteers
The number and severity of treatment emergent adverse events (TEAEs) | 56 days after multiple dose
  To assess the safety and tolerability of multiple oral dose of HSK31858 in healthy volunteers

SECONDARY OUTCOMES:
Cmax | within 30 minutes before administration until 72 hours after administration
  Maximum concentration
Tmax | within 30 minutes before administration until 72 hours after administration
  Time to maximum concentration
AUC0-last | within 30 minutes before administration until until 72 hours after administration
  Area under the drug concentration-time curve, from time 0h to 72h
t½ | within 30 minutes before administration until 72 hours after administration
  Apparent terminal half-life
Absolute neutrophil count (ANC) normalized relative neutrophil elastase (NE) Activity | within 30 minutes before administration until until 56 days after administration
  Assessed NE activity changes in multiple doses

CONTACTS AND LOCATIONS:
Overall Officials: Jie Hou, Principal Investigator — Peking University Care Luzhong Hospital; Hong Wang, Principal Investigator — Peking University Care Luzhong Hospital
Locations (1):
- PKUCare Luzhong Hospital, Zibo, Shang Dong, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Wang Y, Yu C, Hu M, Wang L, Chen M, Liu H, Wu N, Hou J. Safety, tolerability, pharmacokinetics and pharmacodynamics of HSK31858, a novel oral dipeptidyl peptidase-1 inhibitor, in healthy volunteers: An integrated phase 1, randomized, double-blind, placebo-controlled, single- and multiple-ascending dose study. Br J Clin Pharmacol. 2025 Aug;91(8):2262-2272. doi: 10.1002/bcp.70027. Epub 2025 Apr 2. PMID 40170587